CLINICAL TRIAL: NCT01272674
Title: Adiponectin Promotes the Migration of Circulating Progenitor Cells Through p38-mediated Induction of the CXCR4 Receptor
Brief Title: Adiponectin and Circulating Progenitor Cells (CPC) Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: German Research Foundation (Other); Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. A. Linke, Co-investigator, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: adipo2008
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- exercise training (Active Comparator): 4 weeks of supervised physical exercise training
  Interventions: Other: exercise training
- control (No Intervention): sedentary lifestyle
- healthy control (No Intervention)

INTERVENTIONS:
Other: exercise training — 4 weeks supervised physical exercise training
  Arms: exercise training

SUMMARY:
Adiponectin and exercise training contribute to the maintenance of a normal vascular tone by influencing vascular NO bioavailability and concentration and function of endothelial progenitor cells. The molecular mechanisms are only partially understood. Therefore, aim of the present study is to elucidate the effects of Adiponectin on endothelial progenitor cell migration and the underlying signaling pathways. Furthermore, the impact of exercise training on adiponectin-mediated endothelial progenitor cell migration will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* ≤ 75 years of age
* stable coronary artery disease
* preserved left ventricular function
* physical work capacity of ≥ 50
* successful elective percutaneous coronary intervention at study begin

Exclusion Criteria:

* diabetes mellitus
* hypercholesterolemia
* untreated hypertension
* smoking
* myocardial infarction within the last 4 weeks
* significant stenosis of the left main coronary artery

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
migratory capacity of endothelial progenitor cells towards an SDF-1 gradient | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Axel Linke, MD, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (1):
- University of Leipzig, Heart Center, Leipzig, Germany